CLINICAL TRIAL: NCT00606749
Title: A Phase 2 Open-Label Uncontrolled Pilot Study of KC706 in Patients With Stable, Active Pemphigus Vulgaris
Brief Title: Use of KC706 for the Treatment of Pemphigus Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kemia, Inc (Industry)
Responsible Party: Michael R Hodges, MD, Kemia,Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC706-C08
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KC706 — 300 mg once daily (QD) for 12 weeks.

SUMMARY:
The purpose of this study is to determine whether KC706 is effective in the prevention and healing of blisters in patients with pemphigus vulgaris, while the patient remains on stable doses of corticosteroids and/or immunosuppressants.

DETAILED DESCRIPTION:
The present study is designed to follow-up on pre-clinical observations that administration of KC706 is associated with prevention of the development of lesions in a mouse model of PV. Patients participating in this study will be those with active disease in spite of ongoing treatment with corticosteroids and/or immunosuppressive agents. The dose chosen for this clinical study is 300 mg once daily. The primary assessment of interest will be pemphigus lesion status during dosing with KC706.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Diagnosis of pemphigus vulgaris
* Patients must be taking and require either corticosteroid therapy or immunosuppressive therapy or both;
* Immunosuppressive therapy, if any,should have been administered at a stable dose for at least 60 days prior to the Baseline Visit and be well-tolerated, without the expectation that there will be a need to increase that dose during the next 30 days;
* Corticosteroids, if any, should have been administered at a stable dose for at least 30 days prior to the Baseline Visit without expectation that there will be a need to increase that dose during the next 30 days;
* Patients should have active PV skin, scalp or mucosal lesions that meet at least one of the following criteria at the Baseline Visit:

  * > 3 new lesions/week every week in the previous 3 weeks (skin, scalp, and/or mucosal), with healing occurring at a rate to match the appearance of new lesions; or
  * At least 3 active, established lesions with a Pemphigus Lesion Score of at least 2; skin or scalp lesions must be ≥ 5mm in diameter to qualify; there is no size requirement for mucosal lesions; or,
  * 1 large active established skin, scalp, or mucosal lesion > 10 mm;
* Accessibility to veins suitable for venipuncture;
* Patients must be cooperative, able to read, understand and give informed consent, and able to adhere to the study visit schedule and protocol requirements; and,
* Patients must be willing to follow adequate contraceptive measures during the study (both sexes).

Exclusion Criteria:

* Any history of opportunistic infections within 3 months prior to receiving study drug;
* Infection with HIV;
* Past or present diagnosis of hepatitis confirmed by serology or elevated hepatic enzymes;
* History of alcoholic liver disease or cirrhosis;
* Clinically significant concurrent medical disease or laboratory abnormalities evidenced by one or more of the following:

  * Hepatobiliary AST or ALT ≥ 1.5 × upper limit of normal (ULN);alkaline phosphatase ≥ 1.5 × ULN; or, total bilirubin > 90% of the ULN;
  * Renal serum creatinine > 1.5 mg/dL; or, significant proteinuria > 2+ on urinary dip test;
  * Hematologic hemoglobin < 11 mg/dL; leukocytes < 3.5 × 109/L; neutrophils < 1.5 × 109/L; or, platelets < 100 × 109/L;
* Presence or history of malignancy;
* Uncontrolled diabetes (defined as diabetes requiring hospitalization or emergency care in the 3 months prior to first dose of study drug);
* History or suspicion of Gilbert's syndrome;
* Significant blood loss (> 500 mL) within 28 days prior to receipt of study drug;
* Use of an investigational drug within 30 days of screening, or longer if that drug is expected to have long-acting effects (e.g., modulation of B-cell activity);
* Use of Rituximab within the past 6 months;
* Use of intravenous IgG within the past 3 months,
* Current or recent history (within 12 months of screening) of drug or substance abuse, including alcohol;
* Known or suspected pregnancy; nursing mothers;
* Clinically significant abnormality on the screening physical examination performed at the Baseline Visit, laboratory testing, vital signs or electrocardiogram suggestive of significant unstable medical condition other than the disease under study;
* Condition which, in the opinion of the Investigator, could interfere with participation in the study or would put the patient at unacceptable risk;
* History of noncompliance with medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of KC706 to prevent the appearance of new lesions and heal existing lesions, while maintaining stable doses of corticosteroids and/or immunosuppressants in patients with pemphigus vulgaris. | 16 weeks

SECONDARY OUTCOMES:
Evaluate the safety of KC706 in patients with PV and to assess plasma levels of KC706 with once daily dosing. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Werth, MD, Principal Investigator — University of Pennsylvania; Bruce Strober, MD, Principal Investigator — NYU MEDICAL CENTER; Francisco Kerdel, MD, Principal Investigator — Florida Academic Dermatology Centers; Michael Kolodney, MD, Principal Investigator — University of California, Los Angeles; Neil Korman, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Amit Pandya, MD, Principal Investigator — University of Texas Southwestern Medical Center; David Rubenstein, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Victoria Werth, MD, Philadelphia, Pennsylvania, United States